CLINICAL TRIAL: NCT01297023
Title: The Effect of Vitamin D3 Alone and in Combination With Calcium Phosphate on Bone Metabolism in Healthy Adults
Brief Title: Human Intervention Study With Calcium Phosphate and Vitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H47-11
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Subjects
Keywords: calcium phosphate; vitamin d3; bone metabolism; human study
MeSH Terms: interventions — calcium phosphate; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- calcium phosphate (Experimental)
  Interventions: Dietary Supplement: calcium phosphate
- vitamin d (Experimental)
  Interventions: Dietary Supplement: vitamin d
- calcium phosphate and vitamin d (Experimental)
  Interventions: Dietary Supplement: calcium phosphate and vitamin d
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: calcium phosphate — 20 subjects consume for 8 weeks a bread enriched with calcium phosphate [1g calcium/d]
  Arms: calcium phosphate
Dietary Supplement: vitamin d — 20 subjects consume for 8 weeks a bread with vitamin d3 [10µg/d]
  Arms: vitamin d
Dietary Supplement: calcium phosphate and vitamin d — 20 subjects consume for 8 weeks a bread enriched with calcium phosphate [1g calcium/d] and vitamin d3 (10µg/d]
  Arms: calcium phosphate and vitamin d
Other: placebo — All participants consume two weeks before intervention a bread without calcium an vitamin d.
  Arms: placebo

SUMMARY:
The study was conducted to investigate the effect of vitamin d3 alone and in combination with calcium phosphate on bone metabolism and further physiological parameters in healthy subjects. It is postulated that calcium phosphate beneficially influences the bone specific action of vitamin d3.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* pregnancy, lactation
* intake of dietary supplements

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
bone resorption and bone formation markers in blood and urine | 8 weeks

SECONDARY OUTCOMES:
concentration of minerals in blood, stool and urine | 8 weeks
blood lipids | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich-Schiller-University Jena, Institute of Nutrition, Department of Nutritional Physiology
Locations (1):
- Friedrich-Schiller-University Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Trautvetter U, Neef N, Leiterer M, Kiehntopf M, Kratzsch J, Jahreis G. Effect of calcium phosphate and vitamin D(3) supplementation on bone remodelling and metabolism of calcium, phosphorus, magnesium and iron. Nutr J. 2014 Jan 17;13:6. doi: 10.1186/1475-2891-13-6. PMID 24438153